CLINICAL TRIAL: NCT03235063
Title: Registry of Pregnancy Follow-up in Patients With Dilated Cardiomyopathy
Brief Title: Pregnancy and Dilated Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Prog/10/17
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated cardiomyopathy; registry; heart failure; pregnancy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: routinely care- no intervention — routinely care- no intervention

SUMMARY:
Increasing cases of women with dilated cardiomyopathy with a project of pregnancy are observed. However there is few knowledge and publications about cardiac diseases in pregnant women. Moreover the majority of medical articles deal with women with congenital heart diseases, valvular pathologies or peripartum cardiomyopathies, and few data are available in literature about women with dilated cardiomyopathy diagnosed before or during the first months of the pregnancy.

Cardiologist and obstetrician advices are considerably limited when patients with dilated cardiomyopathy have a pregnancy project. Knowledges and know-how are currently based on limited personal experiment or on few clinical cases descriptions.

Pregnancy represents a high-risk situation for patients with dilated cardiomyopathy. Creation of a cohort of pregnant women with dilated cardiomyopathy collecting specific data will allow to have a better overview and to appreciate possibilities of a pregnancy project, evolution risks and modalities for medical attention and to improve follow-up and advices delivered to these patients.

DETAILED DESCRIPTION:
This study is a national (20 centres) retrospective (10 years) and prospective registry of pregnant women with dilated cardiomyopathy.

As this study is observational, medical attention of the enrolled patients will not be modified. No specific visit is planned for the study.

Before the enrolment of the patient, the investigator provides the subject with clear and precise information about the protocol and requests her for written informed consent. The French ethical committee gave the investigators the possibility to include women in the registry if the investigators are unable to inform her (deceased women, no follow-up).

The main objective of the study is to evaluate clinical characteristics and study maternal and neonatal evolution and complications during pregnancy using analysis of the morbi-mortality and clinical and para clinical criteria.

The following data will be compiled in a case report form (e-CRF):

* Risk factors, cardiac history
* BNP or NTproBNP value, echocardiographic data (LVEF and LV diameter)
* Medical treatment before and during the pregnancy
* complications; occurrences during the pregnancy
* Modalities of medical attention during delivery: mother/child Patient's data are coded, and therefore anonymous, by using the inclusion number and initials of the patient (first letter of name and first letter of surname (ex: 01-X_X).

In this prospective and retrospective, multi-centre, clinical study, all patients enrolled in the cohort will be included in the statistical analysis. As an observational non-randomized single arm evaluation, the statistical analyses will be descriptive. A minimum of 100 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of majority
* Followed-up for non-ischemic left heart failure, diagnosed before or during the pregnancy or with peripartum history, with a left ventricular ejection fraction < 50% and/or a left ventricle diameter > 27 mm/m2
* In New York Heart Association (NYHA) class 1 to 4
* Pregnant or with pregnancy history
* Patients with left ventricular non-compaction, valvular cardiomyopathy operated or not can also be enrolled

Exclusion Criteria:

* Refusal for participation
* Ischemic, hypertrophic, restrictive and congenital cardiomyopathies

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: pregnant women with dilated cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
evaluate clinical characteristics | Jan 2018
  Purpose is to realise a French cohort of pregnancies in patients with dilated cardiomyopathy to evaluate clinical characteristics, study maternal and neonatal evolution and complications during pregnancy.
study maternal | Jan 2018
  Purpose is to realise a French cohort of pregnancies in patients with dilated cardiomyopathy to evaluate clinical characteristics, study maternal and neonatal evolution and complications during pregnancy.
neonatal evolution | Jan 2018
  Purpose is to realise a French cohort of pregnancies in patients with dilated cardiomyopathy to evaluate clinical characteristics, study maternal and neonatal evolution and complications during pregnancy.
complications during pregnancy | Jan 2018
  Purpose is to realise a French cohort of pregnancies in patients with dilated cardiomyopathy to evaluate clinical characteristics, study maternal and neonatal evolution and complications during pregnancy.

SECONDARY OUTCOMES:
quarterly blood rate of Brain Natriuretic Peptide (BNP) | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
quarterly blood rate of N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
quarterly evolution of left ventricular ejection fraction | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
left ventricular ejection diameter | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
treatment before and during the pregnancy | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
modalities of medical attention during delivery | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
modalities of mother medical attention during peripartum | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention
modalities of new-born medical attention | Jan 2018
  Analyse specific data of the pregnancy follow-up such as quarterly blood rate of Brain Natriuretic Peptide (BNP) or N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) and cardiac echography for quarterly evolution of left ventricular ejection fraction and diameter measurement Analyse treatment before and during the pregnancy Analyse modalities of medical attention during delivery Analyse modalities of mother medical attention during peripartum Analyse modalities of new-born medical attention

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Noel TROCHU, pu-ph, Principal Investigator — Nantes University Hospital
Locations (15):
- France (15):
  - Chu Angers, Angers
  - Chru de Brest, Brest
  - Hospital Henri Mondor, Créteil
  - Chru Lille, Lille
  - AP-HM, Marseille
  - Chu Nancy, Nancy
  - CHU de NANTES, Nantes
  - CHU NICE, Nice
  - Hospital Salpetrière, Paris
  - Hegp Pompidou, Paris
  - Hospital Lariboisière, Paris
  - Ap-Hp Bichat, Paris
  - Chu Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Toulouse, Toulouse